CLINICAL TRIAL: NCT02159456
Title: Continuous Versus Intermittent Enteral Feeding in Critically Ill Patients: a Prospective, Randomized Controlled Trial
Brief Title: Continuous Versus Intermittent Enteral Feeding in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: feed520
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Nutrition Disorders
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous enteral feeding (Experimental): Continuous enteral feeding via infusion pump is applied for at least 7 days after the start of enteral feeding
  Interventions: Other: Continuous enteral feeding via infusion pump
- Intermittent enteral feeding (Active Comparator): Intermittent enteral feeding via gravity-based infusion is applied for at least 7 days after the start of enteral feeding.
  Interventions: Other: Intermittent enteral feeding via gravity-based infusion

INTERVENTIONS:
Other: Continuous enteral feeding via infusion pump
  Arms: Continuous enteral feeding
Other: Intermittent enteral feeding via gravity-based infusion
  Arms: Intermittent enteral feeding

SUMMARY:
1. Nutritional support during critical illness is important to improve the clinical outcome of patients. Recently, the apply of early enteral nutrition is recommend in critically ill patients on basis of data that enteral nutrition can be helpful to prevent the hospital-acquired infections.

   * However, in critically ill patients, the smooth progress of nutritional support is often hindered by gastrointestinal intolerance, underlying clinical condition, and temporal necessity of procedure or operation.
   * Continuous feeding method, compared with intermittent feeding, is expected to reduce the risk of gastrointestinal intolerance, and improve the nutritional support, but this hypothesis is not supported by appropriate evidences.
2. We will elucidate to compare the efficacy and safety of the continuous feeding method in critically ill patients, compared with the intermittent feeding method.

   * Prospective, randomized controlled study
   * Primary outcome: the achievement rate of target nutritional goal within 7 days after the start of enteral nutrition
   * Secondary outcome: gastrointestinal tolerance, In-ICU/hospital mortality, frequency of hospital-acquired infection, ICU/hospital length-of-stay, duration of mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* adult patient admitted in the intensive care unit
* age 20 years old or more
* The enteral nutritional support is expected to be available within 48 hours after ICU admission

Exclusion Criteria:

* previous abdominal surgery within 1 month
* gastrointestinal bleeding, bowel obstruction, refractory vomiting/diarrhea
* hypersensitivity to prokinetics, history of seizure or phechromocytoma
* enteral feeding via enterostomy or gastrostomy
* difficulty to insert or maintain nasogastric tube
* need for specialized feeding (ex: hemodialysis diet, chronic renal failure diet, diabetes diet)
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-05; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Achievement rate of target nutritional goal | Within 7 days after the start of enteral feeding

SECONDARY OUTCOMES:
Gastrointestinal tolerance | Within 7 days after start of enteral feeding
ICU/hospital mortality | During hospital admission
Frequency of hospital-aquired infection | During hospital admission
ICU/hospital length-of-stay | During hospital admission
Duration of mechanical ventilation | During hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Daehak-ro, Jongno-gu, South Korea